CLINICAL TRIAL: NCT01849718
Title: Nacadia Effect Study - Studying the Effect of Garden Therapy in Relations to People Suffering From Stress
Brief Title: Nacadia Effect Study (NEST)
Acronym: NEST
Status: Completed | Type: Observational
Sponsor: Anne Dahl Refshauge (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor-Investigator, Anne Dahl Refshauge, Phd, Assistant Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Other Study IDs: NEST-704171
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Stress-related Problem

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CBT - Cognitive Behavioural Therapy: 40 participants will receive cognitive behavioural therapy in a clinical setting.
  The duration of the individual sessions are one hour, and there are 1-2 sessions per. week, totaling 20 hours, incl. 4 hours of transition conversations.
  The conversations will be exclusively CBT-based. Number of hours for conversational therapy: 20 hours of individual psychotherapy
- Nacadia Therapy: 40 participants will receive garden therapy in a designed, natural environment.
  The individual sessions last three hours with two sessions per week the first and last week and three sessions per week in week 2-9. This gives a total of 96 hours, including 4 x 3 hours transition conversation and 10 x ½ hour individual interviews.
  Experiences and activities related to the garden environment are integrated with mindfulness exercises. The individual conversations in the Nacadia-therapy will be mindfulness-based CBT.
  10 x ½ an hour of individual psychotherapy.

SUMMARY:
This research project deals with stress treatment in the form of garden therapy in the therapy garden Nacadia. The therapy Garden Nacadia has an evidence-based design that is specially designed for the treatment of stressed people.

Nacadia-therapy can be described as a process in which the patient's health and well-being is assumed to enhance by the presence of the natural environment and through participating in meaningful gardening activities.

NEST concerns research on the effect of Nacadia-therapy. The study consists of randomized and longitudinal studies of the effects of Nacadia-therapy compared to acknowledged cognitive behavioral therapy (CBT).

The outcome measures for example consist of: ability to return to work, health care use, psychological measurements related to stress, health, quality of life and changes in medication use. Further, exploratory studies of the garden therapy in the form of observations and interviews will be performed, to get a better understanding of the garden and the garden activities' importance for the therapeutic purposes.

Hypothesis:

- garden therapy, in a designed natural environment, will lead to improved health and well-being for people who are off sick with stress-related disorders

DETAILED DESCRIPTION:
In order to strengthen the project's quality as evidence-based research, the intervention is designed as a randomized controlled trial comparing two treatments on repeated measurements of the same variables over a period of time.

The treatment options in this study is Nacadia-therapy (garden therapy) and cognitive behavioral therapy (CBT - control group). Because the Nacadia-therapy uses a large number of hours, it has been decided to compare it with the longest conventional treatment that can be offered through the public health insurance of stress-related disorders such as anxiety and depression.

1. Number of participants (N): 80

   1. 40 (n) Nacadia Therapy
   2. 40 (n) CBT
2. Type of environment

   1. The therapy garden Nacadia (outdoors or greenhouse)
   2. Clinic (indoors)
3. Therapists and staff

   1. 2 psychologists and a gardener
   2. 2 psychologists
4. Length of treatment

   1. 10 weeks
   2. 10 weeks
5. Treatment content

   1. 96 hours of Nacadia-therapy (including 79 hours of gardening therapy, 10x½ hour individual conversations, and 4x3 hours of transition conversation)
   2. 20 hours individual CBT (including 16 hours of treating conversational therapy and 4x1 hour of transition conversation)
6. Treatment set-up

   1. Group of 8
   2. Individual

Consistent factors in the two treatment options:

* The psychologists involved in both therapy types are authorized, and trained in CBT.
* Conversational therapy: Psychotherapeutic conversations in both treatments are primarily based on CBT.
* The treatments have the same length of time of 10 weeks

Diverging factors in the two treatment options:

* Environment: In the Nacadia-therapy the treatment is taking place in a designed natural environment, and in CBT the treatment takes place in the psychologists' treatment rooms.
* The number of hours: In Nacadia-therapy the individual sessions last three hours, with two sessions per week the first and last week and three sessions a week in week 2-9. This gives a total of 96 hours, including 4 x 3 hours transition conversation and 10 x ½ hour individual interviews. In CBT, the duration of the individual sessions are one hour, and there are 1-2 sessions per. week, totaling 20 hours, incl. 4 hours of transition conversations.
* Treatment content: in Nacadia-therapy experiences and activities related to the garden environment are integrated with mindfulness exercises. The individual conversations in the Nacadia-therapy will be mindfulness-based CBT, whereas in the control group the conversations will be exclusively CBT-based.
* Number of hours for conversational therapy: 20 hours of individual psychotherapy in CBT, 10 x ½ an hour for individual psychotherapy in Nacadia-therapy.

The project is targeted at citizens who are severely burdened by stress (including ICD categories, F 43.0-9(minus 1 = PTSD), and F45.3), which can be expected to correspond to 6-24 months sick leave.

Data Collection will be carried out through questionnaire surveys (at the beginning and ending of the treatment, and 3, 6, and 12 months after the treatment) as well as as well as from National Data Registers on use of Health care, medicine, and on amount of sick leave. This data will be retrieved three years before treatment and one year after treatment.

ELIGIBILITY:
Inclusion Criteria:

* that they suffer from prolonged stress, and have been on sick leave for that reason in ½ -2 years
* There is no other significant and untreated physical illness behind the symptoms
* There is no other significant and untreated mental illness behind the symptoms, such as personality disorders, bipolar disorders, psychosis or a high degree of sociophobia

Exclusion Criteria:

* Suicidal tendencies or abuse problems

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The project has agreed with a number of surrounding municipalities that they refer participants of both genders who are 20-60 years of age to the project through the rehabilitation institutions 'Incita' and 'Væksthuset', WHO are external collaborators Affiliated with the local job centers. Furthermore, local citizens can through their own doctor / psychiatrist or if they are customers at the Insurance Company 'TopDanmark', join the project. They will be provided with detailed information about the project, the target group and the triage procedure.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Patient-related outcomes - quality of life | One year

SECONDARY OUTCOMES:
Function and health - symptom relief | One year
Health economic evaluation - Cost efficiency (cost-effectiveness) | One year
  1. Lower consumption of health care
  2. Resumption of work
Patient-related outcome (quality of life) | One year
  1. Cost utility
  2. Quality adjusted life years

OTHER OUTCOMES:
Nature consumption | One year
  Specifically for the garden therapy, the participants' nature consumption is a primary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ulrika K Stigsdotter, Professor, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Stigsdotter UK, Corazon SS, Sidenius U, Nyed PK, Larsen HB, Fjorback LO. Efficacy of nature-based therapy for individuals with stress-related illnesses: randomised controlled trial. Br J Psychiatry. 2018 Jul;213(1):404-411. doi: 10.1192/bjp.2018.2. Epub 2018 May 25. PMID 29793558